CLINICAL TRIAL: NCT05472662
Title: A Single-dose, Randomised, Double-blind, Controlled, 2-way Cross-over Study to Assess the Potential for Bronchoconstriction of the New Propellant HFA-152a Versus the Marketed HFA-134a Propellant, in Adult Subjects With Mild Asthma
Brief Title: A Study to Compare the Effects of Two Propellants in Adults With Mild Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CLI-05993AB6-07
Record Dates: First submitted 2022-07-14; First posted 2022-07-25 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): Placebo HFA-152a propellant via pressurised metered-dose inhaler (pMDI):
  Administration: Single-dose administration.
  Interventions: Drug: Placebo 152a
- Reference (Placebo Comparator): Placebo HFA-134a propellant via pressurised metered-dose inhaler (pMDI):
  Administration: Single-dose administration.
  Interventions: Drug: Placebo 134a

INTERVENTIONS:
Drug: Placebo 152a — Placebo pressurised metered-dose inhaler (pMDI) formulated with the 152a propellant
  Arms: Test
Drug: Placebo 134a — Placebo pressurised metered-dose inhaler (pMDI) formulated with the 134a propellant
  Arms: Reference

SUMMARY:
This is a Phase IIa, multicentre, single dose, randomised, double blind, controlled, 2 way cross-over study to evaluate the potential for bronchoconstriction of the new HFA-152a propellant (single dose) versus the marketed HFA-134a propellant (single dose) in adults with mild asthma.

HFA=Hydrofluoroalkane

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any study related procedure.
2. Gender and age: Male or female adults aged from 18 to 75 years old (inclusive).
3. Diagnosis of asthma: documented established diagnosis of mild asthma for at least 6 months according to Step 1 of the Global Initiative for Asthma (GINA) 2021 guidelines.
4. Lung function: subjects with a pre-bronchodilator forced expiratory volume in 1 second (FEV1) ≥60% of the predicted normal value and ≥1.5 L at screening and prior to randomisation, after appropriate wash-out from bronchodilators.
5. Documented excessive variability in lung function.
6. Current asthma therapy: as needed low-dose inhaled corticosteroids (ICS)-formoterol, as needed short-acting β2-agonists (SABA), or low-dose ICS whenever SABA was taken taken not more than twice a week (2 events) in the 4 weeks prior to screening or in the 6 weeks prior to randomisation.
7. Asthma control: controlled or partly controlled based on an Asthma Control Questionnaire© (ACQ-5) score <1.5 at screening and prior to randomisation.
8. Ability to use the inhalers.
9. Ability to comply with the protocol. 10: Female subjects of non-childbearing potential (defined as physiologically incapable of becoming pregnant (i.e. postmenopausal or permanently sterile) and Female subjects of childbearing potential, who accepts the use of highly effective contraceptive methods during the study or with non-fertile male partners.

11. Male subjects fulfilling one of the following criteria:

1. Fertile male subjects with pregnant or non-pregnant women of childbearing potential (WOCBP) partners: they must be willing to use male condom from the signature of the Informed Consent Form (ICF) and until the follow-up visit/call, or;
2. Non-fertile male subjects (contraception is not required in this case), or;
3. Fertile male subjects with women of non-childbearing potential (WONCBP) partner (contraception is not required in this case).

   Exclusion criteria:
   1. History of "at risk" asthma.
   2. Recent exacerbation.
   3. Asthma requiring use of biologics.
   4. Respiratory disorders other than asthma.
   5. Lung cancer or history of lung cancer.
   6. Lung resection.
   7. Lower respiratory tract infection.
   8. Documented coronavirus disease 2019 (COVID-19) diagnosis.
   9. Smoking status: current smoker, or ex-smoker with a smoking history of ≥10 pack-years.
   10. Cancer or history of cancer (other than lung cancer);subject with active cancer or a history of cancer with less than 5 years disease-free survival time.
   11. Cardiovascular diseases: subjects who have known and clinically significant (CS) cardiovascular conditions.
   12. Electrocardiogram (ECG) criteria: any CS abnormal 12-lead ECG that, in the Investigator's opinion, would affect safety evaluations or place the subject at risk.
   13. Central nervous system disorders: subjects with a history of symptoms or significant neurological disease.
   14. Other concurrent diseases: subjects with historical or current evidence of uncontrolled concurrent disease such as, but not limited to, hyperthyroidism, diabetes mellitus or other endocrine disease, haematological disease, autoimmune disorders (e.g. rheumatoid arthritis), gastrointestinal disorders (e.g. poorly controlled peptic ulcer, gastroesophageal reflux disease), significant renal impairment or other disease or condition that might, in the judgement of the Investigator, place the subject at undue risk or potentially compromise the results or interpretations of the study.
   15. Laboratory abnormalities: subjects with CS laboratory abnormalities indicating a significant or unstable concomitant disease.
   16. Alcohol/drug abuse.
   17. Participation to investigational trial: subjects who have received any investigational drug within the 30 days (60 days for biologics) prior to screening.

   16. Hypersensitivity: history of hypersensitivity to any of the study medications components.

   17.Subjects mentally or legally incapacitated. 18. Recent eye surgery or any condition where raised intracranial pressure (caused by forceful exhalation) would be harmful.

   19. For female subjects only: pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until termination of the gestation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — Medicines Evaluation Unit
Locations (1):
- Medicine Evaluation Unit Limited, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- HFA-152a Followed by HFA-134a: HFA-152a and HFA-134a propellant via pressurised metered-dose inhaler (pMDI):
  Administration: Single-dose administration.
  Placebo HFA-152a and Placebo HFA-134a: Placebo pMDI formulated with the propellant HFA-152a/ HFA-134a.
  In this study arm, HFA-152a was used during period 1 and HFA-134a was used during period 2.
- HFA-134a Followed by HFA-152a: HFA-134a and HFA-152a propellant via pressurised metered-dose inhaler (pMDI):
  Administration: Single-dose administration.
  Placebo HFA-134a and Placebo HFA-152a: Placebo pMDI formulated with the propellant HFA-134a/HFA-152a.
  In this study arm, HFA-134a was used during period 1 and HFA-152a was used during period 2.
Period: Overall Study
Arm/Group | HFA-152a Followed by HFA-134a | HFA-134a Followed by HFA-152a
Started | 14 | 11
Completed | 14 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HFA-152a Followed by HFA-134a | HFA-134a Followed by HFA-152a | Total
Number analyzed (Participants) | 14 | 11 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (16.1) | 38.9 (13.3) | 42.0 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 9 | 6 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 14 | 11 | 25
Height [Mean (Standard Deviation); unit: cm] | 171.22 (7.82) | 171.70 (8.34) | 171.43 (7.89)
Weight [Mean (Standard Deviation); unit: kg] | 84.25 (13.34) | 77.11 (10.47) | 81.11 (12.46)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.74 (4.22) | 26.17 (3.08) | 27.61 (3.91)
Smoking status at screening [Count of Participants; unit: Participants]
  Non-smoker | 12 | 7 | 19
  Ex-smoker | 2 | 4 | 6
Duration of smoking [Mean (Full Range); unit: years] | 3.5 [2 to 5] | 5.3 [2 to 8] | 4.7 [2 to 8]
Number of pack-years [Mean (Full Range); unit: pack-years] — Pack years smoked: multiply the number of packs smoked per day by the number of years smoked
  pack-years | 2.00 [1.0 to 3.0] | 1.58 [0.1 to 4.0] | 1.72 [0.1 to 4.0]
Time since first asthma diagnosis [Mean (Full Range); unit: years] | 33.50 [9.6 to 63.6] | 29.41 [21.7 to 43.6] | 31.70 [9.6 to 63.6]
Asthma medication at study entry [Count of Participants; unit: Participants]
  As needed short-acting β2-agonists (SABA) | 12 | 11 | 23
  Low-dose inhaled corticosteroids (ICS) whenever SABA was taken | 2 | 0 | 2
Number of exacerbations in the previous 12 months [Mean (Full Range); unit: Number of exacerbations] | 0.14 [0.0 to 1.0] | 0.00 [0.0 to 0.0] | 0.08 [0.0 to 1.0]
Number of participants with exacerbations (0 or 1) in the previous 12 months, [Count of Participants; unit: Participants]
  0 (no exacerbation) | 12 | 11 | 23
  1 (one exacerbation) | 2 | 0 | 2
Time since the last exacerbation [Mean (Full Range); unit: months] — Population: This item presents data on the time since the last exacerbation (in months) and takes into account duration of longer than 12 months since the last exacerbation. Only participants with available date of the last exacerbation were considered.
  months
    number analyzed (Participants) | 5 | 1 | 6
    (all) | 194.03 [1.7 to 488.4] | 212.40 [212.40 to 212.40] | 197.09 [1.7 to 488.4]
Asthma Control Questionnaire 5 (ACQ-5) total score at screening [Mean (Full Range); unit: score] — The Asthma Control Questionnaire 5 (ACQ-5) is a self-administered questionnaire which includes five questions on asthma symptoms experienced during the past week. Subjects had to score each of the questions on a scale of zero to six, where zero = excellent control of the symptom and six = extremely poor control. The overall score of the ACQ-5 was the mean of the five responses. Subjects had to have an overall score of <1.5 to be eligible for inclusion in this study (inclusion criterion).
  score | 0.43 [0.0 to 1.4] | 0.38 [0.0 to 1.2] | 0.41 [0.0 to 1.4]
Asthma Control Questionnaire 5 (ACQ-5) total score on Day 1, pre-dose [Mean (Full Range); unit: score] — The Asthma Control Questionnaire 5 (ACQ-5) is a self-administered questionnaire which includes five questions on asthma symptoms experienced during the past week. Subjects had to score each of the questions on a scale of zero to six, where zero = excellent control of the symptom and six = extremely poor control. The overall score of the ACQ-5 was the mean of the five responses. Subjects had to have an overall score of <1.5 to be eligible for inclusion in this study (inclusion criterion).
  score | 0.33 [0.0 to 1.0] | 0.29 [0.0 to 0.6] | 0.31 [0.0 to 1.0]

OUTCOME MEASURES:

1. Primary Outcome: Safety: Relative Change From Baseline* in Forced Expiratory Volume in 1 s (FEV1) -- 15 Min Post-dose
Description: Safety: Relative change from baseline* in forced expiratory volume in 1 s (FEV1) at the 15 min post-dose time point. Results are presented as adjusted mean and 95% confidence interval (CI.)
  The potential of the test propellant (HFA-152a vs HFA-134a) for bronchoconstriction was evaluated using centralised spirometry assessments performed during treatment period 1 (TP1) and treatment period 2 (TP2).
  T0 was defined as the moment when the first inhalation took place, and was used to calculate the pre-dose time points.
  T1 was defined as the moment when the last inhalation took place, and was used to calculate the post-dose time points.
  *The baseline FEV1 values were the mean of the two pre-dose assessments (i.e., performed at 45 min and 15 min before T0).
Time Frame: At 15 min post-dose after T1.
Population: Safety set was used: includes all subjects who were randomised and received at least one dose of study drug (HFA-152a or HFA-134a).
Measure: Mean (95% Confidence Interval); unit: percent change
Groups:
- Test: Placebo HFA-152a propellant via pMDI:
  Administration: Single-dose administration.
  Placebo 152a: Placebo pMDI formulated with the 152a propellant
- Reference: Placebo HFA-134a propellant via pMDI:
  Administration: Single-dose administration.
  Placebo 134a: Placebo pMDI formulated with the 134a propellant
Arm/Group | Test | Reference
Number analyzed (Participants) | 25 | 24
percent change | 2.12 [0.52 to 3.72] | 0.26 [-1.37 to 1.89]
Statistical Analysis 1: Comparison: Test vs Reference; Statistical analysis performed on the data at 15 min post-dose timepoint. Statistical analysis was performed by means of Analysis of Covariance (ANCOVA) model including treatment group, subject, and period as fixed effects and FEV1 baseline as covariate; Test type: Equivalence — Equivalence was demonstrated if the 95% CI of the adjusted mean difference in relative change from baseline in FEV1 between HFA-152a and HFA-134a was within the equivalence limits [-10% ; +10%]; p = 0.113, ANCOVA; Adjusted mean difference = 1.86, 95% CI 2-sided [-0.48 to 4.20]

2. Secondary Outcome: Safety: Safety: Relative Change From Baseline* in FEV1 -- All Other Post-dose Time Points
Description: Safety: Relative change from baseline* in FEV1 at all the other post-dose time points (5 min, 30 min, 1 h, 1 h 30 min, and 3 h after T1). Results are presented as adjusted mean and 95% CI.
  The potential of the test propellant (HFA-152a vs HFA-134a) for bronchoconstriction was evaluated using centralised spirometry assessments performed during treatment period 1 (TP1) and treatment period 2 (TP2).
  T0 was defined as the moment when the first inhalation took place, and was used to calculate the pre-dose time points.
  T1 was defined as the moment when the last inhalation took place, and was used to calculate the post-dose time points.
  *The baseline FEV1 values were the mean of the two pre-dose assessments (i.e., performed at 45 min and 15 min before T0).
Time Frame: At 5 min, 30 min, 1 h, 1 h 30 min, and 3 h after T1.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Test | Reference
Number analyzed (Participants) | 25 | 25
percent change
  5 min post-dose: number analyzed (Participants) | 25 | 23
  5 min post-dose | 0.25 [-0.85 to 1.35] | -0.32 [-1.55 to 0.90]
  30 min post-dose | 1.73 [0.57 to 2.89] | 1.50 [0.34 to 2.67]
  1 h post-dose | 1.32 [0.23 to 2.41] | 1.72 [0.63 to 2.81]
  1.5 h post-dose | 2.73 [1.96 to 3.51] | 2.86 [2.09 to 3.64]
  3 h post-dose | 1.91 [0.98 to 2.83] | 2.59 [1.67 to 3.52]
Statistical Analysis 1: Comparison: Test vs Reference; Statistical analysis performed on the data at 5 min post-dose timepoint. Statistical analysis was performed by means of Analysis of Covariance (ANCOVA) model including treatment group, subject, and period as fixed effects and FEV1 baseline as covariate; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.483, ANCOVA; Adjusted mean difference = 0.58, 95% CI 2-sided [-1.10 to 2.25]
Statistical Analysis 2: Comparison: Test vs Reference; Statistical analysis performed on the data at 30 min post-dose timepoint. Statistical analysis was performed by means of Analysis of Covariance (ANCOVA) model including treatment group, subject, and period as fixed effects and FEV1 baseline as covariate; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.782, ANCOVA; Adjusted mean difference = 0.23, 95% CI 2-sided [-1.45 to 1.90]
Statistical Analysis 3: Comparison: Test vs Reference; Statistical analysis performed on the data at 1 h post-dose timepoint. Statistical analysis was performed by means of Analysis of Covariance (ANCOVA) model including treatment group, subject, and period as fixed effects and FEV1 baseline as covariate; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.599, ANCOVA; Adjusted mean difference = -0.40, 95% CI 2-sided [-1.97 to 1.16]
Statistical Analysis 4: Comparison: Test vs Reference; Statistical analysis performed on the data at 1.5 h post-dose timepoint. Statistical analysis was performed by means of Analysis of Covariance (ANCOVA) model including treatment group, subject, and period as fixed effects and FEV1 baseline as covariate; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.815, ANCOVA; Adjusted mean difference = -0.13, 95% CI 2-sided [-1.24 to 0.99]
Statistical Analysis 5: Comparison: Test vs Reference; Statistical analysis performed on the data at 3 h post-dose timepoint. Statistical analysis was performed by means of Analysis of Covariance (ANCOVA) model including treatment group, subject, and period as fixed effects and FEV1 baseline as covariate; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.294, ANCOVA; Adjusted mean difference = -0.69, 95% CI 2-sided [-2.01 to 0.64]

3. Secondary Outcome: Safety: Absolute Change From Baseline* in FEV1 -- All Time Points Post Dose
Description: Safety: Absolute change from baseline* in FEV1 at all post-dose time points. Results are presented as adjusted mean and 95% CI.
  The potential of the test propellant (HFA-152a vs HFA-134a) for bronchoconstriction was evaluated using centralised spirometry assessments performed during treatment period 1 (TP1) and treatment period 2 (TP2).
  T0 was defined as the moment when the first inhalation took place, and was used to calculate the pre-dose time points.
  T1 was defined as the moment when the last inhalation took place, and was used to calculate the post-dose time points.
  The baseline FEV1 values were the mean of the two pre-dose assessments (i.e., performed at 45 min and 15 min before T0).
Time Frame: At 5 min, 15 min, 30 min, 1 h, 1 h 30 min, and 3 h after T1.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Liter
Arm/Group | Test | Reference
Number analyzed (Participants) | 25 | 25
Liter
  5 min post-dose: number analyzed (Participants) | 25 | 23
  5 min post-dose | 0.008 [-0.022 to 0.038] | -0.006 [-0.040 to 0.027]
  15 min post-dose: number analyzed (Participants) | 25 | 24
  15 min post-dose | 0.066 [0.018 to 0.114] | 0.005 [-0.043 to 0.054]
  30 min post-dose | 0.054 [0.019 to 0.088] | 0.049 [0.015 to 0.084]
  1 h post-dose | 0.045 [0.012 to 0.078] | 0.056 [0.023 to 0.089]
  1.5 h post-dose | 0.087 [0.063 to 0.111] | 0.090 [0.066 to 0.114]
  3 h post-dose | 0.059 [0.028 to 0.090] | 0.082 [0.051 to 0.113]
Statistical Analysis 1: Comparison: Test vs Reference; Statistical analysis performed on the data at 5 min post-dose timepoint. Statistical analysis was performed by means of Analysis of Covariance (ANCOVA) model including treatment group, subject and period as fixed effects and FEV1 baseline as covariate; Test type: Other; p = 0.519, ANCOVA; Adjusted mean difference = 0.015, 95% CI 2-sided [-0.032 to 0.061]; Assess differences between treatment groups
Statistical Analysis 2: Comparison: Test vs Reference; Statistical analysis performed on the data at 15 min post-dose timepoint. Statistical analysis was performed by means of Analysis of Covariance (ANCOVA) model including treatment group, subject and period as fixed effects and FEV1 baseline as covariate; Test type: Other; p = 0.085, ANCOVA; Adjusted mean difference = 0.061, 95% CI 2-sided [-0.009 to 0.130]; Assess differences between treatment groups
Statistical Analysis 3: Comparison: Test vs Reference; Statistical analysis performed on the data at 30 min post-dose timepoint. Statistical analysis was performed by means of Analysis of Covariance (ANCOVA) model including treatment group, subject and period as fixed effects and FEV1 baseline as covariate; Test type: Other; p = 0.858, ANCOVA; Adjusted mean difference = 0.004, 95% CI 2-sided [-0.045 to 0.054]; Assess differences between treatment groups
Statistical Analysis 4: Comparison: Test vs Reference; Statistical analysis performed on the data at 1 h post-dose timepoint. Statistical analysis was performed by means of Analysis of Covariance (ANCOVA) model including treatment group, subject and period as fixed effects and FEV1 baseline as covariate; Test type: Other; p = 0.632, ANCOVA; Adjusted mean difference = -0.011, 95% CI 2-sided [-0.058 to 0.036]; Assess differences between treatment groups
Statistical Analysis 5: Comparison: Test vs Reference; Statistical analysis performed on the data at 1.5 h post-dose timepoint. Statistical analysis was performed by means of Analysis of Covariance (ANCOVA) model including treatment group, subject and period as fixed effects and FEV1 baseline as covariate; Test type: Other; p = 0.846, ANCOVA; Adjusted mean difference = -0.003, 95% CI 2-sided [-0.038 to 0.031]; Assess differences between treatment groups
Statistical Analysis 6: Comparison: Test vs Reference; Statistical analysis performed on the data at 3 h post-dose timepoint. Statistical analysis was performed by means of Analysis of Covariance (ANCOVA) model including treatment group, subject and period as fixed effects and FEV1 baseline as covariate; Test type: Other; p = 0.282, ANCOVA; Adjusted mean difference = -0.024, 95% CI 2-sided [-0.068 to 0.021]; Assess differences between treatment groups

4. Secondary Outcome: Safety: Subjects With a Relative Change From Baseline* in FEV1 <-15% -- All Post-dose Time Points
Description: Safety: Number and percentage of subjects with a relative change from baseline* in FEV1 at each post-dose time point <-15%.
  The baseline FEV1 values were the mean of the two pre-dose assessments (i.e., performed at 45 min and 15 min before T0).
Time Frame: At 5 min, 15 min, 30 min, 1 h, 1 h 30 min, and 3 h after T1.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Test | Reference
Number analyzed (Participants) | 25 | 25
Participants
  5 min post-dose | 0 | 0
  15 min post-dose | 0 | 0
  30 min post-dose | 0 | 0
  1 h post-dose | 0 | 0
  1 h 30 min post-dose | 0 | 0
  3 h post-dose | 0 | 0

5. Secondary Outcome: Safety: Change From Baseline* in FEV1 Area Under the Concentration-time Curve From Time Zero to 3 Hours (AUC0-3h)
Description: Change from baseline* in FEV1 area under the concentration-time curve from time zero to 3 hours (AUC0-3h). Results show the change from baseline in FEV1 AUC(0-3h) corrected for Time, in litres
  The potential of the test propellant (HFA-152a vs HFA-134a) for bronchoconstriction was evaluated using centralised spirometry assessments performed during treatment period 1 (TP1) and treatment period 2 (TP2).
  T0 was defined as the moment when the first inhalation took place, and was used to calculate the pre-dose time points.
  T1 was defined as the moment when the last inhalation took place, and was used to calculate the post-dose time points.
  *The baseline FEV1 values were the mean of the two pre-dose assessments (i.e., performed at 45 min and 15 min before T0).
Time Frame: At 3 h post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Test | Reference
Number analyzed (Participants) | 25 | 25
Litres | 0.055 (0.088) | 0.068 (0.081)

6. Secondary Outcome: Safety: Relative Change From Baseline* in Peak Expiratory Flow (PEF) -- All Post-dose Time Points
Description: Safety: Relative change from baseline* in peak expiratory flow (PEF) at all post-dose time points.
  The potential of the test propellant (HFA-152a vs HFA-134a) for bronchoconstriction was evaluated using centralised spirometry assessments performed during treatment period 1 (TP1) and treatment period 2 (TP2).
  T0 was defined as the moment when the first inhalation took place, and was used to calculate the pre-dose time points.
  T1 was defined as the moment when the last inhalation took place, and was used to calculate the post-dose time points.
  The baseline PEF values were the mean of the two pre-dose assessments (i.e., performed at 45 min and 15 min before T0).
Time Frame: At 5 min, 15 min, 30 min, 1 h, 1 h 30 min, and 3 h after T1.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Test | Reference
Number analyzed (Participants) | 25 | 25
percent change
  5 min post-dose: number analyzed (Participants) | 25 | 23
  5 min post-dose | -1.85 (3.74) | -2.35 (3.69)
  15 min post-dose: number analyzed (Participants) | 25 | 24
  15 min post-dose | -0.62 (4.31) | -2.64 (4.35)
  30 min post-dose | -0.19 (3.88) | -0.28 (3.20)
  1 h post-dose | -0.12 (3.95) | 0.11 (4.82)
  1 h 30 min post-dose | 1.96 (4.75) | 1.14 (5.43)
  3 h post-dose | 1.08 (3.57) | 1.62 (4.77)

7. Secondary Outcome: Safety: Absolute Change From Baseline* in PEF -- All Post-dose Time Points
Description: Safety: Absolute change from baseline* in PEF at all post-dose time points. The potential of the test propellant (HFA-152a vs HFA-134a) for bronchoconstriction was evaluated using centralised spirometry assessments performed during treatment period 1 (TP1) and treatment period 2 (TP2).
  T0 was defined as the moment when the first inhalation took place, and was used to calculate the pre-dose time points.
  T1 was defined as the moment when the last inhalation took place, and was used to calculate the post-dose time points.
  The baseline PEF values were the mean of the two pre-dose assessments (i.e., performed at 45 min and 15 min before T0).
Time Frame: At 5 min, 15 min, 30 min, 1 h, 1 h 30 min, and 3 h after T1.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Litres/min
Arm/Group | Test | Reference
Number analyzed (Participants) | 25 | 25
Litres/min
  5 min post-dose: number analyzed (Participants) | 25 | 23
  5 min post-dose | -8.4 (16.5) | -12.5 (20.8)
  15 min post-dose: number analyzed (Participants) | 25 | 24
  15 min post-dose | -2.0 (20.2) | -14.5 (21.5)
  30 min post-dose | -0.8 (20.2) | -2.1 (17.3)
  1 h post-dose | 0.0 (20.0) | -0.3 (24.5)
  1 h 30 min post-dose | 9.9 (23.4) | 3.9 (29.5)
  3 h post-dose | 4.4 (17.9) | 6.5 (24.4)

8. Secondary Outcome: Safety: Subjects With Use of Rescue Medication -- 3 h Post Dose
Description: Number and percentage of subjects with use of rescue medication in the 3 h post dose.
Time Frame: 3 h post-dose.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Test | Reference
Number analyzed (Participants) | 25 | 25
Participants | 0 | 0

9. Secondary Outcome: Safety and Tolerability: Vital Signs -- Diastolic Blood Pressure
Description: Safety and tolerability: Mean change from baseline in the Vital Signs -- Diastolic Blood Pressure
Time Frame: At 45 min, 1.75 h, 2.75 h post dose.
Population: as for outcome 1
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Test | Reference
Number analyzed (Participants) | 25 | 25
mmHg
  Baseline (actual value) | 71.5 [57 to 89] | 72.5 [59 to 87]
  45 min post dose (change from baseline) | 1.4 [-13 to 9] | 0.7 [-14 to 12]
  1.75 h post dose (change from baseline) | 2.8 [-8 to 8] | 1.2 [-15 to 14]
  2.75 h post dose (change from baseline): number analyzed (Participants) | 25 | 24
  2.75 h post dose (change from baseline) | -1.8 [-12 to 9] | -2.7 [-18 to 13]

10. Secondary Outcome: Safety and Tolerability: Vital Signs -- Systolic Blood Pressure
Description: Safety and tolerability: Mean change from baseline in the Vital Signs -- Systolic Blood Pressure
Time Frame: At 45 min, 1.75 h, 2.75 h post dose.
Population: as for outcome 1
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Test | Reference
Number analyzed (Participants) | 25 | 25
mmHg
  Baseline (actual value) | 117.4 [96 to 155] | 115.8 [100 to 135]
  45 min post dose (change from baseline) | 2.3 [-21 to 15] | 1.3 [-16 to 21]
  1.75 h post dose (change from baseline) | 4.9 [-14 to 17] | 2.5 [-9 to 21]
  2.75 h post dose (change from baseline): number analyzed (Participants) | 25 | 24
  2.75 h post dose (change from baseline) | 1.0 [-20 to 13] | 2.0 [-9 to 12]

11. Secondary Outcome: Safety and Tolerability: ECG Parameter -- Heart Rate
Description: Safety and tolerability: Mean change from baseline in the ECG parameter -- Heart rate
Time Frame: At 45 min, 1.75 h, 2.75 h post dose.
Population: as for outcome 1
Measure: Mean (Full Range); unit: beats/min
Arm/Group | Test | Reference
Number analyzed (Participants) | 25 | 25
beats/min
  Baseline (actual value) | 59.4 [45 to 74] | 59.0 [43 to 83]
  45 min post dose (change from baseline) | -3.6 [-19 to 7] | -1.9 [-12 to 11]
  1.75 h post dose (change from baseline) | -3.4 [-15 to 7] | -3.3 [-13 to 6]
  2.75 h post dose (change from baseline) | 5.0 [-6 to 25] | 5.6 [-6 to 13]

12. Secondary Outcome: Safety and Tolerability: ECG Parameter -- PR Interval
Description: Safety and tolerability: Mean change from baseline in the ECG parameter -- PR interval.
Time Frame: At 45 min, 1.75 h, 2.75 h post dose.
Population: as for outcome 1
Measure: Mean (Full Range); unit: msec
Arm/Group | Test | Reference
Number analyzed (Participants) | 25 | 25
msec
  Baseline (actual value) | 154.8 [104 to 203] | 154.2 [99 to 202]
  45 min post dose (change from baseline) | -2.3 [-47 to 8] | 0.4 [-11 to 13]
  1.75 h post dose (change from baseline) | -3.0 [-43 to 15] | -0.9 [-28 to 14]
  2.75 h post dose (change from baseline) | 1.7 [-7 to 22] | -0.3 [-10 to 12]

13. Secondary Outcome: Safety and Tolerability: ECG Parameter -- QRS
Description: Safety and tolerability: Mean change from baseline in the ECG parameter -- QRS interval.
Time Frame: At 45 min, 1.75 h, 2.75 h post dose.
Population: as for outcome 1
Measure: Mean (Full Range); unit: msec
Arm/Group | Test | Reference
Number analyzed (Participants) | 25 | 25
msec
  Baseline (actual value) | 96.6 [77 to 128] | 96.8 [78 to 128]
  45 min post dose (change from baseline) | 0.2 [-9 to 9] | 0.7 [-8 to 10]
  1.75 h post dose (change from baseline) | 1.6 [-8 to 12] | 0.8 [-5 to 12]
  2.75 h post dose (change from baseline) | 1.4 [-11 to 10] | 0.8 [-9 to 9]

14. Secondary Outcome: Safety and Tolerability: ECG Parameter -- QTcF Interval
Description: Safety and tolerability: Mean change from baseline in the ECG parameter -- QTcF interval.
Time Frame: At 45 min, 1.75 h, 2.75 h post dose.
Population: as for outcome 1
Measure: Mean (Full Range); unit: msec
Arm/Group | Test | Reference
Number analyzed (Participants) | 25 | 25
msec
  Baseline (actual value) | 408.4 [380 to 442] | 409.0 [382 to 449]
  45 min post dose (change from baseline) | 0.8 [-14 to 16] | 0.1 [-14 to 18]
  1.75 h post dose (change from baseline) | 4.6 [-12 to 23] | -0.1 [-25 to 18]
  2.75 h post dose (change from baseline) | 5.7 [-11 to 35] | 1.5 [-15 to 19]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were monitored from the screening visit (between 2-21 days before TP1 of the study) to the termination visit, up to 6 weeks.
Description: Safety set was used for the evaluation of AEs.
  Safety set included all subjects who were randomised and received at least one dose of study drug (HFA-152a or HFA-134a).
Arm/Group | Test | Reference
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 1/25 | 3/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (N=25) | Reference (N=25)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators should inform Chiesi Farmaceutici S.p.A. before using the results of the study for publication or presentation, and agree to provide the Sponsor with a copy of the proposed presentation.

DOCUMENTS (2):
  • Study Protocol (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT05472662/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT05472662/SAP_001.pdf